CLINICAL TRIAL: NCT03275714
Title: Evaluation of an App for Smartphones for People With a Bipolar Affective Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: bipolarAPP
Record Dates: First submitted 2017-08-31; First posted 2017-09-07 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Bipolar Affective Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People With a Bipolar Affective Disorder (Active Comparator)
  Interventions: Device: Smartphone APP
- Control subjects without a psychiatric disorder (Active Comparator)
  Interventions: Device: Smartphone APP

INTERVENTIONS:
Device: Smartphone APP — Participants use the BiP-App for 6 months. The app continuously records data on light and motion sensors, as well as Global Positioning System (GPS) and mood surveys.

SUMMARY:
The primary objective of the clinical trial is to evaluate the data of an app for smartphones (BiP-App) with regard to sleep, movement, mood and communication behavior.

The data will be compared between two groups: people with a bipolar affective disorder and individuals without a psychiatric disorder.

Secondary objective of the trial is to investigate if it is possible to detect early warning symptoms of depressive / (hypo) manic episodes via the measured behavior patterns.

Furthermore it will be evaluated whether the BiP-app can find applicability in the examined patient group.

Study design: Clinical evaluation of a medical device without CE mark; Parallel study design

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the participant after clarification
* Patients with a bipolar affective disorder (group of patients) Or control persons without a mental illness (control group)
* Age between 18 and 70 years
* Knowledge about using a smartphone

Exclusion Criteria:

* Rejection of participation
* Lack of knowledge about how to deal with a smartphone
* Congenital / early-childhood intelligence reduction
* Moderate / severe dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Sleep duration | 6 months
  in minutes
Movement behaviour | 6 months
  evaluated through motion sensors and localization services
Mood | 6 months
  evaluated by mood surveys
Communication behaviour | 6 months
  Frequency of usage of communication services

SECONDARY OUTCOMES:
Patient acceptance | 6 months
  evaluated by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für Psychiatrie und Psychotherapeutische Medizin, Graz, Austria